CLINICAL TRIAL: NCT06611592
Title: Safety and Efficacy of Pramipexole Treatment in Resistant Obsessive-Compulsive Disorder (OCD): Pilot, Randomized and Controlled Clinical Trial
Brief Title: Safety and Efficacy of Pramipexole Treatment in Resistant Obsessive-Compulsive Disorder (OCD)
Acronym: OCD-RT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Clinical Academic Center (2CA-Braga) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OCD_rt; 2024-511085-37-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-04; First posted 2024-09-25 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pramipexole at a dose of 0.088 mg/tid (Experimental): Treatment with antidepressant and pramipexole at a dose of 0.088 mg/tid (0.125 mg of salt)
  Interventions: Drug: Pramipexole 0.088mg/tid
- Pramipexole at a dose of 0.18 mg/tid (Experimental): Treatment with antidepressant and pramipexole at a dose of 0.18 mg/tid (0.25 mg of salt)
  Interventions: Drug: Pramipexole 0.18 mg/tid
- Pramipexole at a dose of 0.35 mg/tid (Experimental): Treatment with antidepressant and pramipexole at a dose of 0.35 mg/tid (0.50 mg of salt)
  Interventions: Drug: Pramipexole 0.35 mg/tid

INTERVENTIONS:
Drug: Pramipexole 0.088mg/tid — Week 1 - Week 16 (end of treatment): Oral administration of 0.088 mg/tid dose of pramipexole (0.125 mg of salt).
  Arms: Pramipexole at a dose of 0.088 mg/tid
Drug: Pramipexole 0.18 mg/tid — Week 1: oral administration of 0,088 mg/tid dose of pramipexole (0.125 mg salt).
  Week 2 -Week 16 (end of treatment): oral administration of 0.18 mg/tid dose of pramipexole (0.25 mg salt).
  Arms: Pramipexole at a dose of 0.18 mg/tid
Drug: Pramipexole 0.35 mg/tid — Week 1: oral administration of 0,088 mg/tid dose of pramipexole (0.125 mg salt).
  Week 2: oral administration of a 0.18 mg/tid dose of pramipexole (0.25 mg salt).
  Week 3 - Week 16 (end of treatment): oral administration of a 0.35 mg/tid dose of pramipexole (0.50 mg salt).
  Arms: Pramipexole at a dose of 0.35 mg/tid

SUMMARY:
The most common and effective treatment for OCD is pharmacological therapy that includes selective serotonin reuptake inhibitors (SSRIs) antidepressants and, in the case of patients resistant to this approach, a combination with antipsychotics. Risperidone and aripiprazole are atypical antipsychotics that act on dopamine (D2) and serotonin receptors. Studies have shown that these drugs are effective in boosting SSRIs for the treatment of OCD in resistant patients.

Currently a high percentage of people diagnosed with OCD do not respond to the existing treatments. Pramipexole is a dopaminergic receptor agonist that specifically binds to dopamine D2 and D3 receptors, having demonstrated benefit in resistant depression.

The aim of this clinical trial is to explore how pramipexole can act in the treatment of OCD in resistant patients, evaluating its safety and efficacy.

DETAILED DESCRIPTION:
Phase 2 clinical trial, randomized, with three-parallel-groups, lasting 26 weeks (screening phase, 4 weeks + treatment phase, 16 weeks + follow-up phase, 6 weeks), whose primary objective is to evaluate the effectiveness of using pramipexole as a strategy for boosting SSRIs, in three different doses, in treatment of resistant OCD.

The main endpoint is the measurement of the difference in the total score of the Y-BOCS scale between baseline (V1; before intervention with the investigational drug) and week 16 (V9; after intervention with the investigational drug), between the different groups treated with different doses of pramipexole.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 64 years;
2. European Portuguese as mother tongue;
3. Patients diagnosed with OCD, regardless of subtype, according to DSM-5 and/or ICD-10 criteria;
4. Yale-Brown Obsessive Compulsive Scale (Y-BOCS) score ≥ 16;
5. Patients resistant to the first-line treatment for OCD:

5.1 Patients who do not respond to treatment with at least two selective serotonin reuptake inhibitor antidepressants (SSRIs) at the maximum tolerated therapeutic dose during at least 12 weeks, i.e. patients in whom there is no reduction in the Y-BOCS score by 25% relative to the score obtained before starting treatment with SSRIs.

5.2 Patients who do not respond to treatment with risperidone or aripiprazole as potentiation of the SSRIs at the maximum tolerated therapeutic dose during at least 12 weeks, i.e. patients in whom there is no reduction in the Y-BOCS score by 25% relative to the score obtained before starting treatment with the antipsychotic or patients in whom the Y-BOCS score is kept ≥ 16 after the treatment with the antipsychotic.

Exclusion Criteria:

1. Patients with current or anterior history of psychotic illness (schizophrenia, delusions, among others);
2. Patients with bipolar disorder;
3. Patients with tick disorder;
4. Patients with borderline personality disorder;
5. Patients with social anxiety disorder;
6. Patients with current or anterior history of dietary behavior disorders (at least in the last 6 months);
7. Patients with a history of neurological disease or traumatic brain injury;
8. Patients with history of alcohol abuse or illicit substances (at least in the last 6 months);
9. Patients who are passing or have passed in the last 6 months by a major depressive episode;
10. Patients that undergo deep brain stimulation;
11. Presence of sensory deficits impeding participation in clinical study;
12. Pregnant or in breastfeeding period;
13. Patients who are doing or have done psychotherapy in the last 6 months;
14. Patients doing medication or receiving prohibited treatments;
15. Patients with allergy to pramipexole or any of the excipients;
16. Patients with creatinine clearance ≤ 50 ml/min (calculated by Cockcroft-Gault formula);
17. Patients with NYHA III or IV heart failure or any other severe cardiovascular disease;
18. Hypotension (<90/60 mmHg) sitting position and hypotension orthostatic (drop in systolic AT ≥20 mmHg or diastolic AT ≥10 mmHg after 2-3 minutes of orthostatism) at the screening;
19. Patients with contraindication to perform MRI cannot participate in the assessment of the exploratory endpoint (i.e., other pre-specified outcomes).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2028-08-20 (Estimated); Study Completion 2028-08-20 (Estimated)

PRIMARY OUTCOMES:
Difference between baseline and after treatment in Y-BOCS total score | Baseline and Week 16
  The measurement of the difference in the total score of the Y-BOCS scale between baseline (before intervention with the investigational drug) and after intervention with the investigational drug, between the different groups treated with different doses of pramipexole.
  The Y-BOCS scale measures obsessions separately from compulsions and specifically measures the severity of symptoms of obsessive-compulsive disorder without being biased towards or against the type of content the obsessions or compulsions might present. The final scores range from 0 to 40, with higher scores indicating higher symptom severity. The scores indicate subclinic (0 - 7 points), mild (8 - 15 points), moderate (16 - 23 points), severe (24 - 31 points), and extreme severity (32 - 40 points).

SECONDARY OUTCOMES:
Number of adverse events observed | From Day 2 (after the first dose of the investigational drug) until Week 22 (end of study)
  Number of adverse events observed (nonserious, serious not related to the investigational medicinal product, and serious related to the investigational medicinal product)

OTHER OUTCOMES:
OCI-R Total score | Baseline, Day 1, Day 28, Week 8, Week 12, Week 16, Week 18 and Week 22
  Obsessive-Compulsive Inventory-Revised (OCI-R) is a self-report instrument that assesses the symptoms of OCD during the last month through 18 statements that are related to everyday situations. The total score ranges from 0 to 72 points. Higher scores on this scale indicate higher severity of OCD symptoms.
Scores of the 4 subscales of the WHOQOL-bref | Baseline (before intervention), Week 16 (after intervention ), and Week 22 (end of study)
  The Quality of Life Scale (WHOQOL-bref) is an instrument that assesses four conceptual domains of quality of life: material and physical well-being, relationships with other people, psychological well-being and environment. This self-report instrument, consisting of a brief sociodemographic questionnaire and 26 statements, quantifies global cognitive judgments of life satisfaction.
HAM-D Total score | Baseline, Day 1, Day 7, Day 14, Day 21, Day 28, Week 8, Week 12, Week 16, Week 18 and Week 22
  Hamilton Depression Rating Scale (HAM-D) instrument to measure the psychic and somatic components of depression. From 0 - 7 the participant is considered asymptomatic, while a score equal to or greater than 20 indicates the presence of depressive symptoms. The higher the value, the greater the severity of the symptoms, ranging from moderate to severe.
HAM-A Total score | Baseline, Day 1, Day 7, Day 14, Day 21, Day 28, Week 8, Week 12, Week 16, Week 18 and Week 22
  Hamilton Anxiety Rating Scale (HAM-A) instrument to measure the psychic and somatic components of anxiety. The final scores indicate: mild anxiety (0 - 17 points), moderate anxiety (18 - 24 points) and potentially worrying levels of anxiety (25 - 30 points).
PSS-10 Total score | Baseline, Day 1, Day 28, Week 8, Week 12, Week 16, Week 18 and Week 22
  Perceived Stress Scale (PSS-10) is a self-report questionnaire to assess perceived stress during the last month. The total score can vary between 0 and 40 points. A higher total score indicates higher levels of perceived stress.
SIQ total score | Baseline, Day 1, Day 7, Day 14, Day 21, Day 28, Week 8, Week 12, Week 16, Week 18 and Week 22
  The Suicidal Ideation Questionnaire (SIQ) assesses thoughts and cognitions about suicide and death over the past month. Higher scores in the SIQ scale represent greater severity of suicidal ideation. The total score ranges from 0 to 180 points.
Neurobiological parameters - Cortical thickness | Baseline (before intervention) and Week 16 (after intervention with the investigational drug).
  Anatomical sequence (Magnetization Prepared - RApid Gradient Echo) to assess cortical thickness
Neurobiological parameters - Functional connectivity | Baseline (before intervention) and Week 16 (after intervention with the investigational drug).
  Functional sequences (Echo-planar imaging) at rest to assess functional connectivity of neural networks and static and dynamic connectivity
Neurobiological parameters - Brain activity | Baseline (before intervention) and Week 16 (after intervention with the investigational drug).
  Functional sequences (Echo-planar imaging) during an emotional processing task to assess brain activation during emotional processing
Neurobiological parameters - Diffusion | Baseline (before intervention) and Week 16 (after intervention with the investigational drug).
  Diffusion sequences (Diffusion Weighted Imaging) to measure mean diffusivity (MD), fractional anisotropy (FA), axial diffusivity (AD) and radial diffusivity (RD), in order to assess white matter integrity.
Biochemical parameters - Complete blood count | Baseline (before intervention ), Week 16 (after intervention) and Week 22 (end of the study)
  Blood samples will be collected to measure the complete blood count.
Biochemical parameters - Cortisol | Baseline (before intervention ), Week 16 (after intervention) and Week 22 (end of the study)
  Blood samples will be collected to measure the cortisol.
Biochemical parameters - ACTH | Baseline (before intervention ), Week 16 (after intervention) and Week 22 (end of the study)
  Blood samples will be collected to measure the adrenocorticotropic hormone (ACTH).
Biochemical parameters - T4 | Baseline (before intervention ), Week 16 (after intervention) and Week 22 (end of the study)
  Blood samples will be collected to measure the thyroxine (T4).
Biochemical parameters - TSH | Baseline (before intervention ), Week 16 (after intervention) and Week 22 (end of the study)
  Blood samples will be collected to measure the thyroid stimulating hormone (TSH).
Biochemical parameters - creatinine | Baseline (before intervention ), Week 16 (after intervention) and Week 22 (end of the study)
  Blood samples will be collected to measure the creatinine.
Biochemical parameters - glucose | Baseline (before intervention ), Week 16 (after intervention) and Week 22 (end of the study)
  Blood samples will be collected to measure the glucose.
Biochemical parameters - glycated hemoglobin | Baseline (before intervention ), Week 16 (after intervention) and Week 22 (end of the study)
  Blood samples will be collected to measure the glycated hemoglobin.
Biochemical parameters - Prolactin | Baseline (before intervention ), Week 16 (after intervention) and Week 22 (end of the study)
  Blood samples will be collected to measure the prolactin.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Morgado, MD, PhD, Principal Investigator — 2CA-Braga
Locations (1):
- Clinical Academic Center - Braga (2CA-Braga), Braga, Portugal

IPD SHARING:
Plan to Share IPD: No